CLINICAL TRIAL: NCT05105256
Title: Platelet-rich Plasma Infiltration Versus Corticosteroid Infiltration (Prednisolone) in Treatment of Lumbar Facet Joint Syndrome
Acronym: IAPRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PO21030*
Record Dates: First submitted 2021-10-08; First posted 2021-11-03 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain; Osteoarthritis
MeSH Terms: conditions — Low Back Pain; Osteoarthritis | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The primary and secondary outcomes will be evaluated by a doctor who does not know in which group the patient is randomized.
  This doctor is different from the interventional rheumatologist. Furthermore, the patient is completely unable to determine the group in which he was included. In fact, the infiltrations of the posterior inter-apophyseal joints are carried out in prone position. This technical aspect leads to the patient's ignorance of the treatment received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroids (Active Comparator): Lumbar facet joint injection with corticosteroids
  Interventions: Drug: Prednisolone
- PRP (Experimental): Lumbar facet joint injection with PRP
  Interventions: Drug: Platelet-rich plasma

INTERVENTIONS:
Drug: Prednisolone — Patient will have 1 infiltration of 3mL to 5 mL corticosteroids on average distributed equally over all the posterior joints affected by arthritis phenomena.Lumbar facet joint injection with corticosteroids will be performed at inclusion
  Arms: Corticosteroids
Drug: Platelet-rich plasma — Patient will have 1 infiltration of 3mL to 5 mL of PRP on average distributed equally over all the posterior joints affected by arthritis phenomena.Lumbar facet joint injection with PRP will be performed at inclusion.
  Arms: PRP

SUMMARY:
The prevalence of low back pain is estimated at 90% . Recent studies have shown that 15% to 52% of back pain is attributable to facet joint syndrome .

Being the only vertebral joints provided with a synovial membrane, the posterior inter-apophyseal joints are subject, like all other peripheral joints, to degenerative arthritis phenomena.

These phenomena most often result in the release of pro-inflammatory cytokines resulting in cartilage degradation.

PRP or platelet rich plasma is an autologous blood product obtained after centrifugation of a peripheral blood sample. The PRP has many anti-inflammatory properties. Numerous studies have shown the interest of intra-articular infiltration of PRP in osteoarthritis of the knee but also in tendinopathies of the shoulder and a few studies also suggest the use of PRP in the spine "intra-disc, epidural and posterior joints) .

Corticosteroid infiltrations in the posterior lumbar joints constituting the standard treatment in posterior inter-apophyseal osteoarthritis.

The goal is to obtain a new therapeutic weapon in the management of this frequent and invalid disease for patients who are often elderly and with other comorbidity.

DETAILED DESCRIPTION:
This is a randomized controlled trial, of superiority, which aims to demonstrate that in low back pain induced by osteoarthritis phenomena affecting the facet joint syndrome, PRP infiltrations are greater than that of corticosteroids.

In the context of this study, the patients will have an infiltration of PRP or an infiltration of corticosteroids (the infiltration of corticosteroids corresponds to the usual management of patients with low back pain attributable to posterior inter-apophyseal osteoarthritis).

It has already been shown, in particular in osteoarthritis of the knee that PRP infiltrations do better than local corticosteroid infiltrations at 6 months, with a comparable safety profile.

In low back pain attributable to posterior inter-apophyseal osteoarthritis, the therapeutic possibilities are limited and include either corticosteroid infiltration initially or a surgical intervention.

Corticosteroid injections are the standard treatment, but the maximum limitation of 3 injections per year and the presence of medical contraindications (hypertension, diabetes or uncontrolled infection, etc.) or even operative ones, lead to a therapeutic impasse.

If the investigators show superiority over prednisolone infiltrations, PRP infiltrations may be provided to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient seen at the University Hospital of Reims for an infiltration in the context of pain in low back pain attributable to posterior inter-apophyseal osteoarthritis
* Patient over 18 years old
* Patient presenting at least 5 criteria (and criteria 3) (Cochin criteria):
* Low back pain not exacerbated by cough
* Lumbalgia well relieved by the decubitus
* Low back pain not exacerbated when leaning forward
* Low back pain not exacerbated when getting up
* Low back pain not exacerbated in hyper extension
* Low back pain not exacerbated in Extension - Rotation
* Patient with an MRI dating less than 1 year before inclusion: No herniated disc in the level of the posterior joints to be infiltrated (example: if an infiltration of the post L4-L5 joint is planned, it is considered that there must be no herniated disc at the level L4-L5)
* Patient having signed the consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Contraindications to corticosteroid infiltrations: unbalanced hypertension, unbalanced diabetes, allergy, skin condition next to the infiltration site, not compatible with an infiltration
* Patient who received corticosteroid infiltration within the last 6 months
* Patient who has already received an injection of PRP (for the spine or another indication).
* History of previous spine surgery
* Presence of an ongoing local or systemic infection
* Coagulopathy not compatible with performing a deep gesture
* Pregnant woman and breastfeeding woman
* Presence of motor deficit
* Pain less than 4/10 (ENA)
* Patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
50% improvement in numerical pain scale | 6 months
  50% improvement in ENA (numerical pain scale) without trunk movement at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: No